CLINICAL TRIAL: NCT05157971
Title: A Phase 1 Study Combining Venetoclax With a Pediatric-Inspired Regimen for Newly Diagnosed Adults With B Cell Ph-Like Acute Lymphoblastic Leukemia
Brief Title: Venetoclax and a Pediatric-Inspired Regimen for the Treatment of Newly Diagnosed B Cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21134; NCI-2021-09185 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21134 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: B Acute Lymphoblastic Leukemia; Ph-Like Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Cyclophosphamide; Cytarabine; Daunorubicin; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Prednisone; deltacortene; prednylidene; venetoclax; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (venetoclax, C10403 regimen) (Experimental): See Detailed Description
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisone; Drug: Venetoclax; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given SC, IV or IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pegaspargase — Given IM or IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of venetoclax in combination with a pediatric-inspired chemotherapy regimen known as C10403 in treating patients with newly diagnosed B cell acute lymphoblastic leukemia. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. The C10403 regimen is composed of the chemotherapy drugs cytarabine, cyclophosphamide, daunorubicin, mercaptopurine, pegaspargase, vincristine, and methotrexate, all which work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It also consists of prednisone, which is an anti-inflammatory drug that lowers the body's immune response and is used with other drugs in the treatment of some types of some types of cancer. This study may help researchers learn if adding venetoclax to the pediatric-inspired C10403 regimen can be tolerated and help treat older patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of combining venetoclax with the C10403 regimen backbone during induction and consolidation in newly diagnosed adults with B cell acute lymphoblastic leukemia (ALL).

II. To determine the maximum tolerated dose (MTD) and the recommended phase 2 dose/schedule (RP2D) of venetoclax in combination with the C10403 regimen.

SECONDARY OBJECTIVES:

I. To estimate complete response (CR) after induction. II. To estimate composite CR (CR or CR with incomplete hematologic recovery [CRi] or CR with partial hematologic recovery [CRh]) after induction.

III. To estimate minimal residual disease (MRD) negativity after induction. IV. To estimate MRD negativity after consolidation. V. To estimate CR after induction for Philadelphia (Ph)-like ALL. VI. To estimate CR/CRi/CRh after induction for Ph-like ALL. VII. To estimate MRD negativity after induction for Ph-like ALL. VIII. To estimate MRD negativity after consolidation for Ph-like ALL. IX. To estimate leukemia-free survival (LFS) and overall survival (OS).

OUTLINE:

INDUCTION: Patients receive venetoclax orally (PO) on days 1-14. Patients also receive cytarabine intrathecally (IT) on day 1, prednisone PO twice daily (BID) on days 1-28, vincristine intravenously (IV) on days 1, 8, 15 and 22, daunorubicin IV on days 1, 8, 15 and 22, pegaspargase intramuscularly (IM) or IV on day 4, and methotrexate IT on days 8 and 29 (and also on days 15 and 22 for central nervous system [CNS]3 patients) in the absence of disease progression or unacceptable toxicity. Patients with stable disease (SD) or partial response (PR) after Induction proceed to Extended Induction. Patients with CR, CRi, or CRh after Induction proceed to Consolidation.

EXTENDED INDUCTION: Patients receive venetoclax PO on days 1-7, prednisone PO BID on days 1-14, vincristine IV on days 1 and 8, daunorubicin IV on day 1, and pegaspargase IM or IV on day 4 in the absence of disease progression or unacceptable toxicity. Patients with CR, CRi, or CRh after Extended Induction proceed to Consolidation.

CONSOLIDATION: Patients receive venetoclax PO on days 1-14, cyclophosphamide IV on days 1 and 29, cytarabine IV or subcutaneously (SC) on days 1-4, 8-11, 29-32 and 36-39, mercaptopurine PO on days 1-14 and 29-42, vincristine IV on days 15, 22, 43 and 50, pegaspargase IM or IV on days 15 and 43, and methotrexate IT on days 1, 8, 15 and 22 (omit on days 15 and 22 for CNS3 patients) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age between 18 and 54 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically confirmed B-cell ALL according to World Health Organization criteria

  * Note: Lymphoblastic leukemia is included as long as there is bone marrow involvement
* Newly diagnosed disease with >= 5% blasts in the marrow
* White blood cell count less than 25 x 10^9/L prior to initiation of venetoclax. Cytoreduction with hydroxyurea or steroid or a single dose of intrathecal chemotherapy prior to treatment may be required (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease or underlying leukemia, =< 3 X ULN) (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST) =< 2.5 x ULN (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)

  * Unless it is related to underlying leukemia
* Alanine aminotransferase (ALT) =< 2.5 x ULN (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)

  * Unless it is related to underlying leukemia
* Creatinine clearance of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (performed within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Left ventricular ejection fraction (LVEF) >= 50%

  * Note: Echocardiogram to be performed within 42 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test. (performed within 14 days prior to Day 1 of protocol therapy unless otherwise stated)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control (non-hormonal) or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only

Exclusion Criteria:

* Leukemia-based therapy with chemotherapy with the exception of:

  * Cytoreduction with steroid or hydroxyurea or a single dose of intrathecal chemotherapy is allowed before initiating the study
* Strong or moderate CYP3A4 inducers within 14 days prior to day 1 of protocol therapy
* Subjects who have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Star fruit within 3 days prior to the first dose of study drug
* Live vaccines
* Philadelphia chromosome positive (Ph+; t(9;22)), MLL-rearrangement, t(12;21), and t(1;19)
* T cell ALL
* Class III/IV cardiovascular disability according to the New York Heart Association Classification. Subjects with controlled, asymptomatic atrial fibrillation can enroll
* Parenchymal central nervous system (CNS) involvement requiring cranial radiation
* Participants with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of enrollment
* History of acute cardiovascular ischemic event, i.e., myocardial infarction or unstable angina within 6 months of enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Clinically significant uncontrolled illness
* Uncontrolled active infection
* Other active malignancy
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after completion of treatment
  Will be graded according to the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, frequency, probable association with the study treatment and reversibility or outcome.
Dose limiting toxicity | During cycle 1 (4 weeks)
  Defined as any toxicities that occur during cycle 1, per CTCAE version 5.0, and are considered at least possibly related to venetoclax or the combination of venetoclax and C10403. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, frequency, probable association with the study treatment and reversibility or outcome.

SECONDARY OUTCOMES:
Complete response (CR) after induction +/- extended induction | At week 4 or 6
  Will be estimated and the 95% Clopper Pearson binomial confidence interval (CI) will be estimated.
Complete response (CR) after consolidation | Up to 1 year
  Will be estimated and the 95% Clopper Pearson binomial CI will be estimated.
Composite complete response (CR) (CR/ CR with incomplete hematologic recovery [CRi]/ CR with partial hematologic recovery [CRh]) after induction +/- extended induction | At week 4 or 6
  Will be estimated and the 95% Clopper Pearson binomial CI will be estimated.
Minimal residual disease (MRD) negativity after induction +/- extended induction | At day 28
  Defined as residual leukemia < 0.01% by flow cytometry. Will be estimated and the 95% Clopper Pearson binomial CI will be estimated.
Minimal residual disease (MRD) negativity after consolidation | At week 12
  Will be estimated and the 95% Clopper Pearson binomial CI will be estimated.
Complete response (CR) after induction +/- extended induction for Philadelphia (Ph)-like acute lymphoblastic leukemia (ALL) | At week 4 or 6
  Will be estimated and the 95% Clopper Pearson binomial CI will be estimated.
Complete response (CR) after consolidation for Philadelphia (Ph)-like acute lymphoblastic leukemia (ALL) | Up to 1 year
  Will be estimated and the 95% Clopper Pearson binomial CI will be estimated.
Composite complete response (CR) (CR/ CR with incomplete hematologic recovery [CRi]/ CR with partial hematologic recovery [CRh]) after induction +/- extended induction for Philadelphia (Ph)-like acute lymphoblastic leukemia (ALL) | At week 4 or 6
  Will be estimated and the 95% Clopper Pearson binomial CI will be estimated.
Minimal residual disease (MRD) negativity after induction +/- extended induction for Philadelphia (Ph)-like acute lymphoblastic leukemia (ALL) | At week 4 or 6
  Will be estimated and the 95% Clopper Pearson binomial CI will be estimated.
Minimal residual disease (MRD) negativity after consolidation for Philadelphia (Ph)-like acute lymphoblastic leukemia (ALL) | At week 12
  Will be estimated and the 95% Clopper Pearson binomial CI will be estimated.
Leukemia-free survival | Up to 1 year
  Will be estimated using the Kaplan-Meier product-limit method.
Overall survival | Up to 1 year
  Will be estimated using the Kaplan-Meier product-limit method.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim T Aldoss, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States